CLINICAL TRIAL: NCT06056375
Title: Examining Anti-Racist Healing in Nature to Protect Telomeres of Transitional Age BIPOC for Health Equity
Brief Title: Biological and Behavioral Outcomes of Community Nature Walks
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Charlotte Tate (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Charlotte Tate, Full Professor, San Francisco State University
Organization: San Francisco State University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: X21-013
Record Dates: First submitted 2023-09-14; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Stress, Psychological; Telomere Shortening; Stress Reaction
MeSH Terms: conditions — Stress, Psychological; Fractures, Stress

STUDY DESIGN:
Intervention Model Description: Waitlist control design
Masking Description: Since the study is a waitlisted control, all participants are aware of which condition they are in at any time.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Waitlist Control (Other): Waitlist control; all participants receive the treatment but are in a control condition prior to the treatment
  Interventions: Behavioral: Reclaiming Nature Intervention

INTERVENTIONS:
Behavioral: Reclaiming Nature Intervention — The purpose of the community intervention is to prevent health disparities in Black, Latinx, Pilipinx, and Pacific Islander communities of San Francisco, California.

SUMMARY:
The investigators will test the efficacy of our proposed intervention to reduce embodied stress in four racial/ethnic groups (Black, Latinx, Pilipinx, and Pacific Islander) as a preventative intervention for health disparities found in these communities. The intervention is comprised of two phases. The first consists of community nature walks in a pristine redwood forest for six months. This is followed by chosen nature activities with family and/or friends for three months. The investigators will test the ability of these activities in nature to reduce chronic stress that underpins many health disparities using validated biological, behavioral, and sociocultural measures. The use of these measures is in alignment with the National Institute of Minority Health and Health Disparities (NIMHD) Research Framework, and will increase understanding of individual, interpersonal, community, and social level factors that lead to, and that can eliminate health disparities.

DETAILED DESCRIPTION:
The investigators will test the efficacy of our proposed intervention to reduce embodied stress in four racial/ethnic groups (Black, Latinx, Pilipinx, and Pacific Islander) as a preventative intervention for health disparities found in these communities. The intervention is comprised of two phases. The first consists of community nature walks in a pristine redwood forest for six months. This is followed by chosen nature activities with family and/or friends for three months. The investigators will test the ability of these activities in nature to reduce chronic stress that underpins many health disparities using validated biological, behavioral, and sociocultural measures. The use of these measures is in alignment with the National Institute of Minority Health and Health Disparities (NIMHD) Research Framework, and will increase understanding of individual, interpersonal, community, and social level factors that lead to, and that can eliminate health disparities.

ELIGIBILITY:
Inclusion critieria:

* 18 years or older
* able to commit to a 9-month Nature Intervention (6-month walks; 3-month chosen nature activity)
* spoken languages: English, Spanish, or Tagalog
* able-bodied as in must be able to walk.

Exclusion criteria:

* pregnant women (and other gender identities who are pregnant)
* prisoners
* cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Relative Telomere Length | Baseline (pre-intervention), during intervention, immediate post-intervention, 3 months after intervention
  Relative Telomere Length in the name of the outcome measure.

SECONDARY OUTCOMES:
Hair cortisol concentration | Baseline (pre-intervention), during intervention, immediate post-intervention, 3 months after intervention
  Hair cortisol concentration in the name of the outcome measure.
Self-reported stress (extent of) | Baseline (pre-intervention), during intervention, immediate post-intervention, 3 months after intervention
  Cohen Stress Scale (Likert-type self-reported measurement) in the name of the outcome measure.
Positive mood (extent of) | Baseline (pre-intervention), during intervention, immediate post-intervention, 3 months after intervention
  Positive And Negative Affect Scale International version (PANAS-I) (Likert-type self-reported measurement)

OTHER OUTCOMES:
Steps (number of) | Baseline (pre-intervention), during intervention, immediate post-intervention, 3 months after intervention
  total number of steps per day, assessed by Apple's Health Application on phones in the name of the outcome measure.
Heart rate (average of beats per minute over days) | Baseline (pre-intervention), during intervention, immediate post-intervention, 3 months after intervention
  average beats per minute over days assessed by rate hear application on phones
Sleep quality (extent of) | Baseline (pre-intervention), during intervention, immediate post-intervention, 3 months after intervention
  14-item Sleep Questionnaire (Likert-type self-reported measurement)

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco State University, San Francisco, California, United States